CLINICAL TRIAL: NCT01300377
Title: A DOUBLE-BLIND RANDOMIZED TRIAL ASSESSING THE ASSOCIATION BETWEEN TYPE OF LOCAL ANESTHESIA TREATMENT AND POSTOPERATIVE PAIN IN PATIENTS IN HAVING UNDERGONE ARRHYTHMIA SURGERY
Brief Title: A Trial Assessing The Association Between Type Of Local Anesthesia Treatment And Postoperative Pain In Patients In Having Undergone Arrhythmia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 008-197
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2018-01

CONDITIONS: Post-operative Pain
Keywords: Post-operative pain; pain; pacemaker; defibrillator; post-operative narcotic use; local anesthesia
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine / Lidocaine (Active Comparator): Lidocaine/Bupivacaine mixture - 5cc 1% Lidocaine solution mixed with 5 cc 0.25% Bupivacaine solution administered locally to the surgical site at time of the surgical procedure. Administered once only.
  Interventions: Drug: Bupivacaine / Lidocaine
- Lidocaine (Active Comparator): Lidocaine - 10 cc 1% solution administered locally to the surgical site at time of surgical procedure. Administered once only.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Bupivacaine / Lidocaine — 5cc 1% Lidocaine solution mixed with 5 cc 0.25% Bupivacaine solution administered locally to the surgical site at time of the surgical procedure. Administered once only.
  Arms: Bupivacaine / Lidocaine
Drug: Lidocaine — 10 cc 1% solution administered locally to the surgical site at time of surgical procedure. Administered once only.
  Arms: Lidocaine

SUMMARY:
The goal of the proposed study is to investigate the relationship between two standard treatments, lidocaine or a mixture of lidocaine and bupivacaine, and 1) postoperative pain, and; 2) narcotic use following pacemaker or defibrillator insertion in subjects who undergo arrhythmia surgery at Baylor Heart and Vascular Institute while adjusting for pertinent clinical and/or demographic factors. No control group is necessary.

DETAILED DESCRIPTION:
Patients receiving a pacemaker or defibrillator are currently given Bupivacaine, Lidocaine, or a mixture of the two for local anesthetic treatment (in addition to general anesthesia). The choice of local anesthetic to be used during surgery is based primarily on the differences in time for the anesthetic to take effect and duration thereafter. Lidocaine typically works in less than 1 minute and lasts approximately 45 minutes. Bupivacaine works within 2 to 3 minutes and lasts 4 to 6 hours. Lidocaine is often preferable due to its shorter time of effectiveness. However, its relatively short duration may translate into a higher use of narcotics for pain management during postoperative care - particularly within the first hour following emergence from general anesthesia. Therefore it is conceivable that these patients would have higher levels of pain, higher cost of care related to cost of narcotics, and higher cost of caregiver time required to administer them.

ELIGIBILITY:
Inclusion Criteria:

* Arrythmia patients receiving pacemaker or cardiac defibrillator devices at Baylor Heart and Vascular Institute.

Exclusion Criteria:

* Receiving complicated procedures
* Replacement of parts, not inclusive of leads

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-11; Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 3 Years
  To assess the association between standard local anesthetic choice (Lidocaine or a combination of Marcaine and Lidocaine) and postoperative pain in patients receiving a pacemaker or defibrillator. Pain will be measured using the visual analog scale (a standardized and validated scale) at 3 time points: prior to surgery, once awakened from surgery, and 4 hours after.

SECONDARY OUTCOMES:
Total Post-Operative Narcotic Use | 3 Years
  To assess the association between local anesthetic choice (Lidocaine or a combination of Marcaine and Lidocaine) and narcotic use (including dosages and strength of narcotic) within 4 hours after the patient emerges from general anesthesia. The type, number, and dose of narcotics will be collected up to 4 hours after patient awakens from surgery. Narcotics administered will be standardized to the equivalent dose of morphine.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Jack and Jane Heart and Vascular Institute, Dallas, Texas, United States

DOCUMENTS (2):
  • Informed Consent Form (2012-04-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT01300377/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-06-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT01300377/Prot_SAP_001.pdf